CLINICAL TRIAL: NCT07342296
Title: Induction of Migraine Attacks With Aura Using Pituitary Adenylate Cyclase Activating Polypeptide-38: A Randomized Clinical Trial
Brief Title: Induction of Migraine Attacks With Aura Using Pituitary Adenylate Cyclase Activating Polypeptide-38
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Haidar Al-Khazali, Principal Investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-23042432
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Migraine With Aura; Migraine Aura
Keywords: migraine; aura; Pituitary Adenylate Cyclase Activating Polypeptide-38
MeSH Terms: conditions — Migraine with Aura; Migraine Disorders; Epilepsy | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Intervention Model Description: This single-center trial applies a randomized, double-blind, placebo-controlled, two-way crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pituitary Adenylate Cyclase Activating Polypeptide-38 (PACAP-38) (Experimental): PACAP-38 will be administered by intravenous infusion.
  Interventions: Drug: Pituitary Adenylate Cyclase Activating Polypeptide-38 (PACAP-38)
- Placebo (Placebo Comparator): Placebo (isotonic saline) will be administered by intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pituitary Adenylate Cyclase Activating Polypeptide-38 (PACAP-38) — The participants will receive a continuous intravenous infusion of 10 pmol/kg/min PACAP-38 over 20 min
  Arms: Pituitary Adenylate Cyclase Activating Polypeptide-38 (PACAP-38)
Drug: Placebo — The participants will receive a continuous intravenous infusion of 20 mL of placebo (isotonic saline) over 20 minutes.
  Arms: Placebo

SUMMARY:
Pituitary Adenylate Cyclase Activating Polypeptide-38 (PACAP-38) is a key neuropeptide in migraine pathophysiology and treatment. This study investigates whether PACAP-38 administration can trigger aura in individuals with a diagnosis of migraine with aura.

DETAILED DESCRIPTION:
In a series of studies, pharmacological triggers of migraine headache were able to induce aura as well migraine headache. Recent open-label findings show that calcitonin gene-related peptide (CGRP) can trigger aura attacks-despite its limited ability to cross the blood-brain barrier. This suggests CGRP might induce migraine aura via trigeminovascular activation, the same pathway involved in migraine headache. To further explore this concept, it is fundamental to examine whether other migraine-inducing signaling molecules that pass the BBB to a minimal degree, such as PACAP-38, are able to induce aura as well. If PACAP-38 is able to induce aura, the anti-PACAP monoclonal antibody may provide a promising therapeutic option for preventing migraine with aura.

To validate this effect, a randomized, double-blind, placebo-controlled trial is essential. Its outcomes could inform future therapies targeting the migraine-aura connection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* History of migraine with aura for ≥ 12 months according to the International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria
* ≥ 1 monthly day with aura that meets criteria as aura on average across the three months before screening
* Provision of informed consent prior to initiation of any study-specific activities/procedures.

Exclusion Criteria:

* Any history of a primary or secondary headache disorder other than migraine without aura, migraine with aura, chronic migraine, and episodic tension-type headache
* History or evidence of any other clinically significant disorder, condition, or disease (except for those outlined above) that, in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Initiation, discontinuation, or change of dosing of prophylactic medications within 2 months prior to study inclusion
* Intake of acute medications (e.g. analgesics, triptans) within 48 hours of infusion start
* Headache of any intensity within 48 hours of infusion start
* Aura within 48 hours of infusion start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of migraine attacks with aura | 12 hours
  Difference in incidence of migraine attack with aura between PACAP-38 and placebo during the 12-hour observational period after infusion start.
  Experimentally induced migraine aura is defined as aura that meet Criteria B and C of 1.2 Migraine with Aura in ICHD-3.

SECONDARY OUTCOMES:
Incidence of migraine attacks without aura | 12 hours
  Difference in incidence of migraine pain (headache) between PACAP-38 and placebo during the 12-hour observational period after infusion start.
  Experimentally induced migraine pain is defined as headache that meet Criteria C and D of 1.1. Migraine without Aura in ICHD-3 as well as resembles the subject's usual migraine attack or is treated with an acute headache medication.
Headache intensity scores | 12 hours
  Difference in area under the curve (AUC) for headache intensity scores between PACAP-38 and placebo during the 12-hour observational period after infusion start.
  The intensity of headache is rated by the subject on the 11-point numerical rating scale (0 being no headache, 10 being the worst imaginable headache).

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data not published within this article will be made available on reasonable request from any qualified investigator.